CLINICAL TRIAL: NCT07039890
Title: An Open Label, Balanced, Randomized, Single Dose, Two Treatment, Two Sequence, Two Period, Two Way Crossover, Oral Bioequivalence Study in Healthy, Adult, Human Subjects Under Fasting Condition.
Brief Title: To Compare and Evaluate the Oral Bioavailability of Empagliflozin + Linagliptin 10 mg/5 mg Filmcoated Tablets With That of Glyxambi 10 mg/ 5 mg Film-coated Tablets in Healthy, Adult, Human Subjects Under Fasting Conditions.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 24-VIN-0556
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin + Linagliptin filmcoated tablets (Experimental): Empagliflozin + Linagliptin 10 mg/5 mg filmcoated tablets
  Interventions: Drug: Empagliflozin + Linagliptin filmcoated tablets; Drug: Glyxambi film-coated tablets
- Glyxambi film-coated tablets (Active Comparator): Glyxambi 10 mg/5 mg film-coated tablets
  Interventions: Drug: Empagliflozin + Linagliptin filmcoated tablets; Drug: Glyxambi film-coated tablets

INTERVENTIONS:
Drug: Empagliflozin + Linagliptin filmcoated tablets — Empagliflozin + Linagliptin 10 mg/5 mg filmcoated tablets
Drug: Glyxambi film-coated tablets — Glyxambi 10 mg/5 mg film-coated tablets

SUMMARY:
To compare and evaluate the oral bioavailability of Empagliflozin + Linagliptin 10 mg/5 mg film-coated tablets with that of Glyxambi 10 mg/ 5 mg film-coated tablets in healthy, adult, human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 to 45 years (both inclusive).
* Subjects' weight within normal range according to normal values for Body Mass Index (between 18.5 to 30.0 kg/m2) (both inclusive) with minimum of 45 kg weight.
* Subjects with normal health as determined by personal medical history, clinical examination and laboratory examinations within the clinically acceptable range.
* Subject with Creatinine Clearance ≥80 ml/min.
* Subjects having clinically acceptable 12-lead electrocardiogram (ECG).
* Subjects having clinically acceptable chest X-Ray (PA view), if taken.
* Subjects having negative urine screen for drugs of abuse (including amphetamines, barbiturates, benzodiazepines, marijuana, cocaine, and morphine).
* Subjects having negative urine alcohol test / breath alcohol test.
* Non-smoker.
* Subjects willing to adhere to the protocol requirements and to provide written informed consent.
* For male Subjects:

  •Subjects willing to follow approved birth control methods (a double barrier method) for the duration of the study as judged by the investigator(s), such as (a double barrier method) condom with spermicide, Condom with diaphragm, or abstinence. Subjects willing to refrain from donating sperm during the study period.
* For Female Subjects:

  * Female of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as intrauterine device (IUD), abstinence, bilateral tubal ligation or double barrier contraception, i.e., condom + diaphragm, condom + spermicidal or foam
  * Postmenopausal for at least 1 year, or if less than 1 year, then following acceptable contraceptive measures as mentioned above
* Subjects having negative urine pregnancy test at screening and negative serum β-hCG pregnancy test on admission day of period 01 (only for female subjects).

Exclusion Criteria:

* Hypersensitivity to Empagliflozin & Linagliptin or related class of drugs or any of its excipients or heparin.
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological, urogenital or psychiatric disease or disorder.
* Any treatment which could bring about induction or inhibition of hepatic microsomal enzyme system within 30 days prior to admission in period 01.
* History or presence of alcoholism or drug abuse.
* History of any type of acute metabolic acidosis (such as lactic acidosis, diabetic ketoacidosis).
* History or presence of asthma, urticaria or other significant allergic reactions.
* History or presence of significant gastric and/or duodenal ulceration.
* History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumor.
* History or presence of cancer or basal or squamous cell carcinoma.
* Difficulty with donating blood.
* Difficulty in swallowing solids dosage form like tablets or capsules.
* Use of any prescribed medication or OTC medication including vaccines, vitamins and herbal remedies during last 30 days prior to admission in period 01.
* Major illness within past 3 months.
* Volunteer who have donated blood (1 unit) or participation in a drug research study within past 90 days prior to the first dose of the study drug.
* Consumption of xanthine-containing products, tobacco containing products or alcohol or any alcohol containing products within 48.00 hours prior to admission in period 01.
* Consumption of grapefruit or grapefruit juice containing products within 72.00 hours prior to admission of period 01.
* Positive screening test for any one or more: HIV, Hepatitis B and Hepatitis C.
* History or presence of significant easy bruising or bleeding.
* History or presence of significant recent trauma.
* Subjects who have been on an abnormal diet (for whatever reason) during the four weeks preceding the study.
* History of acute conditions with the potential to alter renal function.
* Female subjects who are currently breast feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-08 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 72 hours
  For Empagliflozin: 80.00%-125.00% for geometric least square mean ratio (T/R) and it's 90% confidence intervals for Cmax
Area Under the Curve from time zero to time of last measurable concentration (AUC0-t) | 72 hours
  For Empagliflozin: 80.00%-125.00% for geometric least square mean ratio (T/R) and it's 90% confidence intervals for AUC0-t
Peak Plasma Concentration (Cmax) | 72 hours
  For Linagliptin: 80.00%-125.00% for geometric least square mean ratio (T/R) and it's 90% confidence intervals for Cmax
Area Under the Curve from time zero to time of last measurable concentration (AUC0-72) | 72 hours
  For Linagliptin: 80.00%-125.00% for geometric least square mean ratio (T/R) and it's 90% confidence intervals for AUC0-72

SECONDARY OUTCOMES:
Area Under the Curve from time zero to time infinite (AUC0-∞) | 72 hours
  For Empaglifozin: Descriptive Statistics
Time to reach peak plasma concentration (Tmax) | 72 hours
  For Empagliflozin: Descriptive Statistics
Time to reach peak plasma concentration (Tmax) | 72 hours
  For Linagliptin: Descriptive Statistics

CONTACTS AND LOCATIONS:
Locations (1):
- Veeda Clinical Research Ltd., Ahmedabad, Gujarat, India